CLINICAL TRIAL: NCT01564940
Title: Human Factors Usability Study of Abbreviated Functional Use of the Intimate Bridge 2 Conception, Inc. Conception System
Brief Title: Human Factors Usability Study of Ib2C Conception System
Status: Completed | Type: Observational
Sponsor: Rinovum Women's Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Ib2C-11-015
Record Dates: First submitted 2012-03-25; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Cervical Cap Insemination
Keywords: Cervical cap insemination; Usability Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to obtain subjective feedback in a home use environment regarding usability and ease of use of the applicator and conception cap and the instructions for use. Data will be collected and evaluation to determine if the usability requirements of the conception system as determined by the usability specification have been met. The study will not involve sexual intercourse or delivery of any fluids to the cervix. The study will only involve use of the applicator to insert the cervical cap into the vagina, track it to the cervix and prepare and release the cervical cap (with removal string attached) onto the cervix. The conception cap will remain in place for no more than 6 hours.

DETAILED DESCRIPTION:
The purpose of this study is to obtain subjective feedback in a home use environment regarding usability and ease of use of the applicator and conception cap and the instructions for use. Data will be collected and evaluation to determine if the usability requirements of the conception system as determined by the usability specification have been met. The study will not involve sexual intercourse or delivery of any fluids to the cervix. The study will only involve use of the applicator to insert the cervical cap into the vagina, track it to the cervix and prepare and release the cervical cap (with removal string attached) onto the cervix. The conception cap will remain in place for no more than 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* Female, any ethnicity
* 20 - 45 years of age
* Sexually active
* Signed Informed Consent

Exclusion Criteria:

* Prior surgery to the cervix or vaginal tract
* Vaginal prolapse
* Cervical cancer
* Hysterectomy
* History of Toxic Shock Syndrome (TSS)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females between the ages of 20 and 45.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Pelekanos, OB-GYN, Principal Investigator — Forbes Regional Hospital (West Penn Allegheny Health System)
Locations (1):
- Forbes Regional Hospital, Monroeville, Pennsylvania, United States